CLINICAL TRIAL: NCT05489588
Title: Evaluation of the GORE® VIAFORT Vascular Stent for Treatment of Symptomatic Iliofemoral Venous Obstruction
Brief Title: The GORE® VIABAHN® FORTEGRA Venous Stent Iliofemoral Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNS 21-07
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboses; Venous Disease; Venous Leg Ulcer; Venous Stasis; Venous Ulcer; Venous Stenosis; Venous Occlusion; Vein Thrombosis; Vein Occlusion; Vein Disease
Keywords: VIAFORT; Vein Stent; Venous Thrombosis; Venous Stenosis; Gore; Venous Occlusion; FORTEGRA; VIABAHN FORTEGRA; Venous Disease; Deep Venous Insufficiency; Venous disease treatment Options; Deep venous; DVT Treatment; Venous Stent; Venous insufficiency treatment options
MeSH Terms: conditions — Venous Thrombosis; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, non-randomized, single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GORE® VIAFORT Vascular Stent (Experimental): GORE® VIAFORT Vascular Stent
  Interventions: Device: GORE® VIAFORT Vascular Stent

INTERVENTIONS:
Device: GORE® VIAFORT Vascular Stent — Treatment of unilateral symptomatic iliofemoral venous obstruction with the GORE® VIAFORT Vascular Stent.

SUMMARY:
This study is a prospective, non-randomized, multicenter, single-arm, clinical study to evaluate the performance, safety and efficacy of the GORE® VIABAHN® FORTEGRA Venous Stent (formerly known as GORE® VIAFORT Vascular Stent) for treatment of symptomatic iliofemoral venous obstruction.

DETAILED DESCRIPTION:
A maximum of 30 clinical sites across the U.S. will participate in the study. One hundred and sixty-five subjects are intended to be implanted with the GORE® VIABAHN® FORTEGRA Venous Stent (formerly known as GORE® VIAFORT Vascular Stent) in this study, with a limit of 33 treated subjects per site. Subjects will be evaluated through hospital discharge and return for follow-up visits at 1, 6, 12, 24, 36, 48, and 60 months post-treatment.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient is willing and able to comply with all follow-up evaluations as well as any required medication or compression regimen.
* Patient is able to provide informed consent.
* One of the following: Clinical severity class of CEAP 'C' classification ≥3 or rVCSS pain score ≥2.
* Intention to treat the target areas with only the GORE® VIAFORT Vascular Stent.
* Estimated life expectancy ≥1 year.
* Patient is ambulatory (use of assistive walking device such as a cane or walker is acceptable).
* Patient has adequate inflow to the target lesion(s), per investigator/sub-investigator discretion, involving at least a patent femoral or deep femoral vein.
* Presence of non-malignant symptomatic unilateral iliofemoral venous obstruction.

Preoperative Exclusion Criteria:

* Patient has DVT in the target areas with symptom onset date greater than 14 days but less than or equal to 90 days prior to treatment.
* Patient is a pregnant or breastfeeding woman, or a woman planning to become pregnant through the 12-month visit.
* Patient has clinically significant (e.g., symptoms of chest pain, hemoptysis, dyspnea, hypoxia, etc.) pulmonary embolism (confirmed via Computed Tomography Angiography) at the time of enrollment.
* Patient has a known uncorrectable bleeding diathesis or active coagulopathy meeting the following definitions (all must be tested for):

  1. uncorrected INR>2 (not as a result of warfarin or DOAC therapy), OR
  2. platelet count <50,000 or >1,000,000 cells/mm3, OR
  3. white blood cell count <3,000 or >12,500 cells/mm3
* Patient has impaired renal function (eGFR <30 mL/min/1.73m2) or is currently on dialysis.
* Patient has uncorrected hemoglobin of <9 g/dL.
* Patient has known history of antiphospholipid syndrome (APS).
* Patient has known homozygous or acquired coagulation defect (e.g., Protein C or Protein S deficiency) that cannot be treated with therapeutic anticoagulation.
* Patient has a planned surgical intervention that has the potential to clinically interfere with the endpoints of this treatment (other than pre-stenting procedures such as thrombolysis or thrombectomy) within 30 days prior to or within 30 days after the planned study procedure. Examples include surgical interventions that may impact mobility, and surgical interventions that require cessation of therapeutic antiplatelet or anticoagulation within 30 days following the index procedure.
* Patient has had or requires open deep venous surgery in the target limb.
* Patient is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this treatment, in the opinion of the investigator/sub-investigator. Observational studies are permitted.
* Patient has had a previous major (i.e., above the ankle) amputation of the target lower limb.
* Patient has known sensitivity to device materials.
* Patient has had prior stenting or grafts in the target vessels.
* Patient has a known or suspected active systemic infection at the time of the index procedure. Patients with a chronic infection (e.g., HIV, hepatitis C) that can be managed, and with an active clinical plan in place may be eligible.
* Patient has known history of intravenous drug abuse within one year of treatment.
* Patient has significant peripheral arterial disease (chronic Rutherford Type 2 or greater, acute Rutherford Type IIa or greater).
* Patient has a BMI >45. Patients with a BMI of up to 45 may be enrolled provided that diagnostic quality ultrasound of the implant sites can be performed.
* Patient is actively undergoing or plans to begin cancer treatment.
* Patients with hypercoagulable states that are unwilling to take anticoagulant medications on a long-term basis.
* Patient has contraindication to thrombolytics, anticoagulants, or iodinated contrast necessary for the index procedure and long-term medical therapy (contrast pre-medication is acceptable).

Intraoperative Inclusion Criteria:

* Presence of non-malignant unilateral obstruction of the common femoral vein, external iliac vein, and/or common iliac vein defined as occlusion or at least 50% reduction in target vessel lumen as measured by procedural IVUS and venogram.
* Patient can accommodate an appropriately sized GORE® VIAFORT Vascular Stent as per reference vessel diameter (see IFU), as determined by intraoperative IVUS post pre-dilation.
* Patient must have appropriate access vessels to accommodate the delivery sheath for the selected device size.
* Patient has adequate landing zones free from significant disease requiring treatment within the native vessels beyond the proximal and distal margins of the lesion.
* Patient has adequate inflow to the target lesion(s), per investigator/sub-investigator discretion, involving at least a patent femoral or deep femoral vein.
* Lesion can be traversed with a guidewire.
* Disease involves only unilateral iliofemoral venous segments with intent to stent all affected iliofemoral segments. Patients with disease extending into the inferior vena cava or contra-lateral iliofemoral veins who are anticipated to require endovascular or surgical treatment within 12 months after investigational device implant will be excluded.
* Patient does not have significant (i.e., >20% residual thrombosis) acute thrombus within the target stent area at the time of investigational device placement. Patients with acute thrombus within the target stent area must have thrombus successfully treated prior to investigational device placement. Successful thrombus treatment is defined as reestablishment of antegrade flow with ≤20% residual thrombosis as confirmed by IVUS and venogram, AND freedom from bleeding, vascular injury, or hemodynamically significant pulmonary embolism. After successful thrombus treatment, investigational device placement can occur within the same procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Composite of safety events | 12 months (Stent Embolization) or 30 days (all other components)
  Composite primary safety endpoint consisting of freedom from the following:
  * Stent embolization through 12-month follow-up
  * Device- or procedure-related death through 30 days
  * Clinically significant pulmonary embolism confirmed via Computed Tomography Angiography through 30 days
  * Device- or procedure-related vascular injury through 30 days requiring surgical or endovascular intervention
  * Device- or procedure-related major bleeding events through 30 day
Primary efficacy as assessed by primary patency | 12 months
  Rate of subjects with primary patency as confirmed by imaging and adverse events

SECONDARY OUTCOMES:
Number of subjects with primary patency as confirmed by imaging and adverse events | 60 months
  Number of subjects with freedom from both:
  * stent occlusion due to restenosis or thrombosis as confirmed with imaging, and
  * clinically driven target lesion revascularization as confirmed with imaging and adverse events
Number of subjects with secondary patency as confirmed by imaging and adverse events | 60 months
  Freedom from permanent loss of blood flow through the device, regardless of reintervention.
Number of subjects with clinically driven target lesion revascularization as confirmed by imaging and adverse events | 60 months
  Number of subjects with repeat endovascular procedures (e.g., PTA, stenting, thrombectomy/thrombolysis) to restore flow, performed within the margins of the investigational devices due to ≥50% restenosis of the target lesion as measured via imaging AND the failure to improve or recurrence of venous origin leg pain or venous edema related to the target lesion present at baseline, or the onset of new symptoms including venous origin pain and venous edema related to the target lesion.
Number of subjects with device fracture as confirmed with imaging | 60 months
  Number of subjects with device fracture as confirmed with imaging.
Number of subjects with stent embolization as confirmed with imaging | 12 months
  Number of subjects with stent embolization as confirmed with imaging
Number of subjects with device- or procedure-related death | 30 days
  Number of subjects with device- or procedure-related death
Number of subjects with clinically significant pulmonary embolism as confirmed with imaging and adverse events | 30 days
  Number of subjects with clinically significant pulmonary embolism confirmed via Computed Tomography Angiography through 30 days.
Number of subjects with device- or procedure-related vascular injury as confirmed with adverse events | 30 days
  Number of subjects with device- or procedure-related vascular injury through 30 days requiring surgical or endovascular intervention.
Number of subjects with device- or procedure-related major bleeding events as confirmed with adverse events | 30 days
  Number of subjects with device- or procedure-related major bleeding events through 30 days.
Revised Venous Clinical Severity Scale (rVCSS) | 60 months
  Change in Revised Venous Clinical Severity Scale (rVCSS) Measurement through 60-month follow-up compared to baseline prior to treatment.
  Note: The rVCSS scale ranges from 0 to 30, with higher scores reflecting worse symptoms.
Revised Venous Clinical Severity Scale (rVCSS) Pain | 60 months
  Change in Revised Venous Clinical Severity Scale (rVCSS) Pain Measurement through 60-month follow-up compared to baseline prior to treatment.
  Note: The rVCSS Pain scale ranges from 0 to 3, with higher scores reflecting worse pain.
Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) VEINES-QOL/Sym | 60 months
  Change in Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) Measurement through 60-month follow-up compared to baseline prior to treatment.
Villalta | 60 months
  Change in Villalta Measurement through 60-month follow-up compared to baseline prior to treatment.
5 Level EuroQol-5 Dimension (EQ-5D-5L) | 60 months
  Change in 5 Level EuroQol-5 Dimension (EQ-5D-5L) Measurement through 60-month follow-up compared to baseline prior to treatment.
Technical success | Index procedure (post-op day 0)
  Number of subjects with successful delivery and deployment of the stent to the intended location, and removal of delivery system.
Lesion success | Index procedure (post-op day 0)
  Number of subjects with evidence of ≤50% residual stenosis at the conclusion of the index procedure as measured by IVUS or venogram.
Procedural success | Index procedure through hospital discharge (discharge estimated as up to 30 days post-treatment)
  Number of subjects with lesion success and the absence of major adverse events (i.e., stent embolization, device- or procedure-related death, clinically significant pulmonary embolism, device- or procedure-related vascular injury requiring surgical or endovascular intervention, and device- or procedure-related major bleeding) prior to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kush Desai, MD, Principal Investigator — Northwestern University; Kathleen Gibson, MD, Principal Investigator — Lake Washington Vascular Surgeons
Locations (27):
- United States (27):
  - Stanford University School of Medicine, Stanford, California
  - Advanced Heart and Vein (ClinRe), Thornton, Colorado
  - Vascular Care Group, Darien, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vascular Care Group, Wellesley, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Englewood Hospital & Med Center, Englewood, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Stony Brook, Stony Brook, New York
  - St. Peter's Vascular Associates, Troy, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health-Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Bethesda North, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - UT Southwestern, Dallas, Texas
  - Sentara General Hospital, Norfolk, Virginia
  - Overlake Hospital, Bellevue, Washington
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No